CLINICAL TRIAL: NCT07369947
Title: The Effect of Watching Artificial-Intelligence-Assisted Breastfeeding Videos on Breastfeeding Self-Efficacy, Motivation, and LATCH Scores in First-Time Mothers: A Randomized Controlled Trial
Brief Title: The Effect of Artificial-Intelligence-Assisted Videos on Breastfeeding Self-Efficacy, Motivation, and LATCH Scores in First-Time Mothers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025/559
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Artificial Intelligence (AI); Motivation; Self Efficacy; Midwifery
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : AI-Assisted Breastfeeding Video Group (Experimental)
  Interventions: Procedure: AI-Assisted Breastfeeding Video
- No Intervention : Control Group (No Intervention)

INTERVENTIONS:
Procedure: AI-Assisted Breastfeeding Video — The intervention consists of an AI-supported relaxing breastfeeding video designed to enhance maternal calmness, confidence, and instinctive breastfeeding perception during the early postpartum period. The video is generated using Kling AI through controlled text-to-video workflows. To ensure ethical safety and cultural sensitivity, the content does not include real human or animal breastfeeding images. Instead, it features abstract and metaphorical visuals (e.g., pastel silhouettes, minimalist line-art, or flat illustrations) symbolizing bonding, rhythm, and closeness. The final version is selected following expert review and pilot testing. The video lasts 10 minutes and includes low-level white noise (<60 dB) to support maternal relaxation and infant comfort. Participants in the intervention group watch the video twice, at the 2nd and 6th postpartum hours, via tablet while breastfeeding in a comfortable position, in addition to standard breastfeeding care.
  Arms: Experimental : AI-Assisted Breastfeeding Video Group

SUMMARY:
As of 2024, nearly half (48%) of infants under six months worldwide are exclusively breastfed, approaching the global target of 50%. Building on this progress, the World Health Organization has extended the target to 60% by 2030, emphasizing the need for innovative, scalable, and supportive interventions to strengthen breastfeeding practices. Breastfeeding has well-established benefits for infant growth, immunity, and long-term health, while also reducing maternal postpartum complications and chronic disease risks. Early postpartum support, particularly within the first hours after birth, is critical for successful and sustained breastfeeding. However, in busy clinical settings, providing continuous and individualized support can be challenging, especially for primiparous women who may experience low confidence, pain, and insufficient guidance. This randomized controlled trial aims to evaluate the effect of an artificial intelligence (AI)-supported relaxing breastfeeding video on breastfeeding self-efficacy, breastfeeding motivation, and LATCH scores among primiparous women. Unlike instructional videos, the AI-based video is designed to promote emotional relaxation, instinctive breastfeeding perception, and maternal confidence during the early postpartum period. The study adopts a two-arm randomized controlled experimental design. The population consists of primiparous women who deliver vaginally at Ağrı Training and Research Hospital postpartum unit between February and June 2026. A priori power analysis (α=0.05, power=0.95) indicated a minimum sample size of 38 participants; considering a 20% attrition rate, a total of 46 women (23 per group) will be recruited. Eligible participants include primiparous, Turkish-speaking women without postpartum or neonatal complications. Women who undergo cesarean delivery, have medical or psychiatric conditions preventing breastfeeding, or whose newborns require intensive care will be excluded. Participants will be randomized into intervention and control groups using an online randomization tool. All participants will receive a standardized 5-minute breastfeeding education based on the Turkish Ministry of Health breastfeeding counseling guidelines. In addition to standard care, the intervention group will watch a 10-minute AI-supported relaxing video at the 2nd and 6th postpartum hours during breastfeeding. The video will be displayed via tablet while the mother is in a comfortable breastfeeding position. The control group will receive standard care only. The AI-generated video will be produced using Kling AI, a generative video platform that enables controlled text-to-video workflows. To ensure ethical and cultural sensitivity, the video will not include real human or animal breastfeeding images. Instead, it will feature abstract, metaphorical visuals (e.g., pastel silhouettes, minimalist line art, or flat illustrations) that convey calmness, bonding, rhythm, and instinctive closeness. The final version will be selected following expert review and pilot testing with three postpartum women. Low-level white noise (<60 dB) will accompany the video to enhance maternal relaxation and infant comfort. Data collection tools include a demographic information form, the Breastfeeding Self-Efficacy Scale-Short Form, the Primipara Breastfeeding Motivation Scale, and the LATCH Breastfeeding Assessment Tool. Breastfeeding observations and LATCH scoring will be conducted by an independent midwife blinded to group allocation. Statistical analyses will include descriptive statistics, paired and between-group comparisons, and repeated-measures analyses where appropriate. Ethical approval will be obtained from the relevant institutional ethics committee, and written informed consent will be secured from all participants. The findings are expected to contribute novel evidence on the role of AI-supported emotional and relaxing digital interventions in enhancing early postpartum breastfeeding outcomes and maternal confidence.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* Single pregnancy
* Vaginal delivery
* No complications during the postpartum period
* No visual or auditory communication problems
* Women who speak and read Turkish.

Exclusion Criteria:

* Women who had a cesarean delivery
* Women with severe psychiatric conditions or impaired consciousness
* Women with conditions preventing breastfeeding (e.g., nipple problems, anatomical absence of the breast)
* Women requiring emergency surgical/medical intervention
* Presence of conditions preventing the newborn from breastfeeding (such as cleft palate/lip)
* Newborn admission to the NICU or presence of serious congenital anomalies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Motivation | Baseline (prior to intervention), 2 hours postpartum, and 6 hours postpartum
  Breastfeeding motivation will be measured using the Primipara Breastfeeding Motivation Scale (PBMS), assessing maternal motivation across four domains: value of breastfeeding, self-efficacy, perceived midwife support, and success expectancy. Higher scores indicate greater breastfeeding motivation. The scale, consisting of 29 items and 29-203 points, is interpreted as indicating that women's motivation to breastfeed increases as their scores increase.
Breastfeeding Self-Efficacy | Baseline (prior to intervention), 2 hours postpartum, and 6 hours postpartum
  Breastfeeding self-efficacy will be assessed using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), a validated 14-item Likert-type scale measuring maternal confidence in breastfeeding behaviors. The lowest possible score on the scale is 14, and the highest possible score is 70. A higher score indicates greater breastfeeding self-efficacy.
Breastfeeding Effectiveness (LATCH Score) | 2 hours postpartum and 6 hours postpartum
  Breastfeeding effectiveness will be evaluated using the LATCH Breastfeeding Assessment Tool, which assesses latch, audible swallowing, nipple type, maternal comfort, and positioning/hold. Each domain is scored from 0 to 2, with total scores ranging from 0 to 10; higher scores indicate more effective breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No